CLINICAL TRIAL: NCT04735146
Title: Co-design and Evaluation of the Feasibility and the Efficacy of a Multiple-targeted Adapted Physical Activity Intervention to Promote Quality of Life, Well-being and Physical Activity Levels in Pregnant Women: the WELL-DONE! Study.
Brief Title: Adapted Physical Activity to Promote Quality of Life, Well-being and Physical Activity Levels in Pregnant Women (WELL-DONE!Study)
Acronym: WELL-DONE!
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Cycle Degree in Midwifery in collaboration with the Department of Biomedical and Neuromotor Sc (Other)
Responsible Party: Principal Investigator, Dila Parma, Master's degree in Nursing and Midwifery Sciences, University of Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 984/2020/Sper/AOUBo
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Pregnant Women

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Experimental Group will be involved in 1 weekly session of adapted physical activity lasting 1 hour for 6 weeks within the normal cycle of accompanying birth meetings provided by the University Hospital of Bologna.
  Interventions: Other: Adapted physical activity
- Control Group (No Intervention): The control group is expected to participate in 6 birth accompaniment meetings held online, 1 hour of which will be dedicated to the topic of exercise and physical activity recommendations in pregnancy.

INTERVENTIONS:
Other: Adapted physical activity — Participants in the experimental group will undergo the adapted physical activity program that will be co-designed during phase I of the study.
  The 6-week program is aimed at improving the quality of life; increase the physical activity levels according to recommended guidelines; improving body awareness through an educational component; maintain and ameliorate the previous functions (for women previously active) and build the exercise background for sedentary women; increase physical fitness and functional capacity.
  Arms: Experimental Group

SUMMARY:
The aim of the WELL-DONE! Study is to co-design, using different professional figures (midwives, psychologists, master's degree in motor science) but also taking into consideration the pregnant women's point of view, an intervention of adapted physical activity for pregnant women, included in the birth accompaniment courses and conducted by midwives, and to evaluate its effectiveness in terms of quality of life, well-being, levels of physical activity and satisfaction with respect to the proposed intervention.

DETAILED DESCRIPTION:
The primary objective is the evaluation of an integrated, co-designed intervention of adapted physical activity, included in the birth accompaniment courses, in order to improve the quality of life of pregnant women.

* The secondary objective is the evaluation of the feasibility, efficacy and safety of the intervention in terms of general satisfaction with the proposed intervention, levels of physical activity practiced, physical performance, self-efficacy, sleep quality, anxiety and depression.
* The tertiary objective is to translate, adapt and validate in Italian a specific questionnaire to measure physical activity levels in pregnant women, Pregnancy Physical Activity Questionnaire (PPAQ), through the use of Actigraph accelerometers (ActiLife6 wGT3X-BT ).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the 24th and 32th week.
* Pregnant women belonging to the birth accompaniment meetings organized by University Hospital of Bologna

Exclusion Criteria:

* Alterations in communication skills and / or sensory functions so severe as to make it impossible to understand and / or execute the instructions given by the trainer (dementia, aphasia, blindness, deafness);

  * Premature Rupture of Membranes (PROM).
  * Premature labor.
  * Vaginal bleeding.
  * Placenta previa after 28 weeks gestation.
  * Pre-eclampsia
  * Cervical incontinence
  * Intrauterine fetal growth delay or arrest.
  * Plurigemellarità
  * Uncontrolled type I diabetes.
  * Uncontrolled hypertension.
  * Uncontrolled thyroid disease.
  * Other severe cardiovascular, respiratory or systemic disorders.
  * Any other condition the operator deems may contraindicate participation in a moderate intensity exercise program.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Women's Quality of Life | Baseline (T1); after 6 weeks of intervention (T2); 3 months after childbirth (T3)
  12-Item Short-Form Health Survey (SF-12 Questionnaire)

SECONDARY OUTCOMES:
Change in Physical activity levels | Baseline (T1); follow-up after 6 weeks (T2); 3 months after childbirth (T3)
  Pregnancy Physical Activity Questionnaire (PPAQ)
Change in Physical Performance | Baseline (T1); after 6 weeks of intervention (T2); 3 months after childbirth (T3)
  Six minutes walking distance; Sit to stand test

CONTACTS AND LOCATIONS:
Overall Officials: Dila Parma, Principal Investigator — University of Bologna, Department of Medical and Surgical Sciences
Locations (1):
- Corso di Laurea in Ostetricia - Scuola di Medicina e Chirurgia Alma Mater Studiorum - Università di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No